CLINICAL TRIAL: NCT03831698
Title: Omega 3 Fatty Acids in Colorectal Cancer (CRC) Prevention in Patients With Lynch Syndrome (COLYNE)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-Omega3-CRC-Prev
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Lynch Syndrome
Keywords: Omega 3
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omega-3, 2 grams (Experimental): Omega-3 fatty acid ethyl esters (2 grams) orally (by mouth) once per day for 12 months
  Interventions: Drug: Omega-3 fatty acid ethyl esters (2 gram)

INTERVENTIONS:
Drug: Omega-3 fatty acid ethyl esters (2 gram) — Omega-3 fatty acid ethyl esters (2 gram)
  Other Names: lovaza

SUMMARY:
This is a pilot study aimed at assessing the effects of moderate dose omega-3-acid ethyl esters capsules (generic Lovaza) on molecular, and intestinal microbiota changes in participants at high risk for colorectal cancer. The study will be a single arm, open label study.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant or Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Candidate for elective endoscopy procedure
* Participants with known Lynch Syndrome
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Willing to undergo a colonoscopy and biopsy at baseline and another colonoscopy and biopsy at 12 months visit.
* Participants taking Aspirin for chemoprevention must agree to stop it for at least 4 weeks prior to study entry and throughout the trial period
* Adequate organ and marrow function
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use two forms of adequate contraception (hormonal AND barrier method of birth control) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately.
* Men of child-bearing potential must not father a child or donate sperm while on this study and for 90 days after their last study treatment.

Exclusion Criteria:

* Current or anticipated use of other investigational agents while participating in this study.
* Psychiatric illness/social situations that could limit compliance with study requirements.
* Pregnant or breast feeding.
* Familial adenomatous polyposis, Putz-Jeghers disease, ulcerative colitis, or Crohn's disease.
* Previous or known active malignancies, except non-melanoma skin cancers, unless curatively treated and with no evidence of recurrence for more than 5 years
* Current use of anticoagulation therapy
* Current use of therapeutic doses of aspirin for reasons other than chemoprevention
* Use of omega 3 fatty acids or flaxseed supplements within 4 weeks before this study's screening/baseline colonoscopy
* Use of high dose omega 3 fatty acids within the past 3 months prior to study baseline/screening
* Current, regular use of non-steroidal anti-inflammatory drugs (NSAIDS)
* Allergy to fish and/or fish products
* Uncontrolled infectious disease
* Malabsorption syndrome, disease affecting gastrointestinal function, or previous resection of the stomach or small bowel.
* Unable to swallow and retain oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Retention rate of participants | 12 months
  Feasibility is defined as at least 80% retention rate

SECONDARY OUTCOMES:
Proportion of participants with treatment-related adverse events in each arm. | 12 months
  Measured by Common Terminology Criteria Adverse Events (CTCAE) V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Anwaar Saeed, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (1):
- The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No